CLINICAL TRIAL: NCT07213479
Title: Feasibility and Acceptability of Remote Home-Based Isometric Exercise and Lifestyle Change for the Management of Hypertension
Brief Title: Feasibility and Acceptability of Isometric Exercise and Lifestyle Change for the Management of Hypertension
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: HealthWorks Newcastle Upon Tyne (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 10198
Record Dates: First submitted 2025-09-04; First posted 2025-10-09 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Hypertension (HTN)
Keywords: Hypertension; Isometric Exercise; Wall Squat; Cardiovascular Disease; Lifestyle Change; Blood Pressure
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Individuals who meet the study criteria and agree to participate will be randomly assigned to one of two parallel groups: (1) home-based isometric exercise and lifestyle advice intervention, or (2) lifestyle advice control group. Randomisation will be performed with minimisation for sex and the mean of 24-hour ambulatory systolic BP (≤140 mm Hg vs >140 mm Hg).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home Based Isometric Exercise and Lifestyle Change Group (Experimental): Participants randomised to this group will undertake a remotely supervised 12-week home-based isometric exercise training intervention 3 times per week. The bilateral leg isometric exercise consists of 5-stage wall squat position determined by individual calculations at baseline. Rate of perceived exertion (RPE) will be monitored throughout the intervention and used to guide the squat stage position. Lifestyle change advice will be given in accordance with NICE guidelines for hypertension. Participants will receive a smartwatch (Huawei D2) to monitor their daily physical activity (step count) and record their home blood pressure.
  Interventions: Behavioral: Isometric Exercise and Lifestyle Change Advice
- Lifestyle Change Control Group (Active Comparator): Participants randomised to this group will not receive any intervention other than lifestyle change advice in accordance with NICE guidelines for hypertension. Participants will receive a smartwatch (Huawei D2) to monitor their daily physical activity (step count) and record their home blood pressure.
  Interventions: Behavioral: Lifestyle Change Advice

INTERVENTIONS:
Behavioral: Isometric Exercise and Lifestyle Change Advice — The intervention consists of two distinct phases:
  • Intensive Phase (12 weeks) - a structured, high-support period involving three weekly supervised isometric exercise sessions and lifestyle change advice. The supervised exercise programme will consist of 4 × 2-minute bouts of wall squat exercise, with 2-minute rest periods between bouts. Participant squat height position will be based on individual calculations determined at baseline. Target rate of perceived exertion (RPE) for each bout will be:
  * Bout 1: RPE 4 (target range: 3.5-4.5)
  * Bout 2: RPE 5.5 (target range: 5-6)
  * Bout 3: RPE 7 (target range: 6.5-7.5)
  * Bout 4: RPE 8.5 (target range: 8-9) If the RPE falls outside the target zone for a given bout, participants will adjust their squat height accordingly.
  Lifestyle change advice will be given in booklet form in accordance with current NICE guidelines for hypertension.
  • Maintenance Phase (12-24 weeks) - focus on sustaining exercise and lifestyle behaviour changes
  Other Names: Static Strength Training; Behaviour Change
  Arms: Home Based Isometric Exercise and Lifestyle Change Group
Behavioral: Lifestyle Change Advice — Lifestyle change advice given as per current standard care for hypertension
  Other Names: Behavioural Change
  Arms: Lifestyle Change Control Group

SUMMARY:
High blood pressure (hypertension) is a leading risk factor for cardiovascular diseases and may contribute to poor health and premature death. The purpose of this research is to learn if a home-based isometric exercise programme combined with lifestyle change advice is a practical and acceptable method for people diagnosed with hypertension to manage their condition. Isometric exercise involves a muscle contraction without movement of the limbs and previous research has shown this may be effective for reducing blood pressure. Therefore, this study will explore the experiences, thoughts, attitudes, and barriers to participation. It will also examine the effect the isometric exercise has on blood pressure.

Participants will undertake an isometric exercise programme using a wall squat position, 3 times per week, for 12 weeks. The exercise sessions will be completed at home with remote online supervision by an exercise professional. Lifestyle change advice will given in line with current guidelines to promote healthy behaviours to reduce high blood pressure. After 12 weeks, participants will be encouraged to continue with the wall squat exercise for a further 12-weeks unsupervised. Throughout the study, participants' blood pressure and daily activity will be recorded using a smartwatch device.

Upon completion of the intervention period, participants will be interviewed to gather their views and opinions on the isometric exercise programme. Changes in blood pressure will be evaluated at 12 and 24 weeks.

By exploring whether an isometric exercise programme is a feasible and acceptable method for hypertensive people to manage their condition and how this influences blood pressure, this research may aid in the development of a strategy to manage hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Arterial Hypertension (AH) in accordance with NICE guidelines.
* Under pharmacological treatment for AH with antihypertensive drug, type and dose maintained for the previous four months.
* Blood Pressure with values <180 and <110 mmHg for office systolic and diastolic BP, respectively.
* Not currently engaged in any structured or supervised exercise training programme, including resistance, aerobic, or isometric exercise, defined as planned exercise performed ≥2 times per week at moderate or greater intensity, for at least three months prior to enrolment.
* Written informed consent provided.

Exclusion Criteria:

* Body mass index >35 kg/m2.
* Presence of cardiovascular disease beyond hypertension.
* Known orthopaedic, musculoskeletal, or neurological conditions that restrain isometric exercise execution.
* Presence of secondary hypertension
* Inability to follow verbal instructions or complete study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-02-02 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Intervention | Baseline to 24 weeks
  Feasibility will be determined by the rate of screening, eligibility, recruitment, and retention at 12 and 24 weeks.
Feasibility of Intervention | Baseline to 24 weeks
  Feasibility will be determined by adherence to the intervention (number of sessions attended and completed)
Acceptability of Intervention | Post 24 weeks
  Participant acceptability will be determined through a qualitative process evaluation involving semi-structured interviews. The interviews will identify action mechanisms, examine experiences, barriers, facilitators, and behaviour change strategies, with a diverse sample to reflect varied demographics. Participants will be asked about their experience of participating in the study, thoughts, and attitudes towards the intervention.

SECONDARY OUTCOMES:
Office and Ambulatory Blood Pressure | Baseline to 24 weeks.
  Blood pressure will be measured in mmHg via office and ambulatory methods. Office BP will be taken in a seated position in accordance with resting BP protocols. Ambulatory BP monitoring will be performed with a non-invasive oscillometric device placed on the nondominant arm and programmed to perform measurements every 15 minutes for 24 hours. The secondary outcome is the change in mmHg for systolic and diastolic blood pressure from baseline, 12 weeks, and 24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Cucato, PhD, Principal Investigator — Northumbria University
Locations (1):
- Northumbria University, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] World Health Organisation (2023). Global report on hypertension: the race against a silent killer. Report No.: ISBN 978-92-4-008106-2. Available from: https://www.who.int/publications/i/item/9789240081062.
- [Background] Whelton PK, Carey RM, Aronow WS, Casey DE Jr, Collins KJ, Dennison Himmelfarb C, DePalma SM, Gidding S, Jamerson KA, Jones DW, MacLaughlin EJ, Muntner P, Ovbiagele B, Smith SC Jr, Spencer CC, Stafford RS, Taler SJ, Thomas RJ, Williams KA Sr, Williamson JD, Wright JT Jr. 2017 ACC/AHA/AAPA/ABC/ACPM/AGS/APhA/ASH/ASPC/NMA/PCNA Guideline for the Prevention, Detection, Evaluation, and Management of High Blood Pressure in Adults: Executive Summary: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Hypertension. 2018 Jun;71(6):1269-1324. doi: 10.1161/HYP.0000000000000066. Epub 2017 Nov 13. No abstract available. PMID 29133354
- [Background] Unger T, Borghi C, Charchar F, Khan NA, Poulter NR, Prabhakaran D, Ramirez A, Schlaich M, Stergiou GS, Tomaszewski M, Wainford RD, Williams B, Schutte AE. 2020 International Society of Hypertension global hypertension practice guidelines. J Hypertens. 2020 Jun;38(6):982-1004. doi: 10.1097/HJH.0000000000002453. No abstract available. PMID 32371787
- [Background] Swift HT, O'Driscoll JM, Coleman DD, Caux A, Wiles JD. Acute cardiac autonomic and haemodynamic responses to leg and arm isometric exercise. Eur J Appl Physiol. 2022 Apr;122(4):975-985. doi: 10.1007/s00421-022-04894-7. Epub 2022 Jan 28. PMID 35089384
- [Background] Maisyaroh A., Putri D A., Abdillah A., & Widianto E P. (2021). The effect of isometric exercise on reducing blood pressure in people with hypertension: A literature review. Nurse and Health: Journal Keperawatan. 10(2): 162 - 174.
- [Background] Mancia G, Kreutz R, Brunstrom M, Burnier M, Grassi G, Januszewicz A, Muiesan ML, Tsioufis K, Agabiti-Rosei E, Algharably EAE, Azizi M, Benetos A, Borghi C, Hitij JB, Cifkova R, Coca A, Cornelissen V, Cruickshank JK, Cunha PG, Danser AHJ, Pinho RM, Delles C, Dominiczak AF, Dorobantu M, Doumas M, Fernandez-Alfonso MS, Halimi JM, Jarai Z, Jelakovic B, Jordan J, Kuznetsova T, Laurent S, Lovic D, Lurbe E, Mahfoud F, Manolis A, Miglinas M, Narkiewicz K, Niiranen T, Palatini P, Parati G, Pathak A, Persu A, Polonia J, Redon J, Sarafidis P, Schmieder R, Spronck B, Stabouli S, Stergiou G, Taddei S, Thomopoulos C, Tomaszewski M, Van de Borne P, Wanner C, Weber T, Williams B, Zhang ZY, Kjeldsen SE. 2023 ESH Guidelines for the management of arterial hypertension The Task Force for the management of arterial hypertension of the European Society of Hypertension: Endorsed by the International Society of Hypertension (ISH) and the European Renal Association (ERA). J Hypertens. 2023 Dec 1;41(12):1874-2071. doi: 10.1097/HJH.0000000000003480. Epub 2023 Sep 26. PMID 37345492
- [Background] Luengo-Fernandez R, Leal J, Gray A, Petersen S, Rayner M. Cost of cardiovascular diseases in the United Kingdom. Heart. 2006 Oct;92(10):1384-9. doi: 10.1136/hrt.2005.072173. Epub 2006 May 15. PMID 16702172
- [Background] Kounoupis A, Papadopoulos S, Galanis N, Dipla K, Zafeiridis A. Are Blood Pressure and Cardiovascular Stress Greater in Isometric or in Dynamic Resistance Exercise? Sports (Basel). 2020 Mar 28;8(4):41. doi: 10.3390/sports8040041. PMID 32231128
- [Background] Jones NR, McCormack T, Constanti M, McManus RJ. Diagnosis and management of hypertension in adults: NICE guideline update 2019. Br J Gen Pract. 2020 Jan 30;70(691):90-91. doi: 10.3399/bjgp20X708053. Print 2020 Feb. No abstract available. PMID 32001477
- [Background] O'Driscoll JM, Giorgione V, Edwards JJ, Wiles JD, Sharma R, Thilaganathan B. Myocardial Mechanics in Hypertensive Disorders of Pregnancy: a Systematic Review and Meta-Analysis. Hypertension. 2022 Feb;79(2):391-398. doi: 10.1161/HYPERTENSIONAHA.121.18123. Epub 2021 Nov 17. PMID 35020458
- [Background] Bytyci Katanolli A, Probst-Hensch N, Ann Obas K, Gerold J, Zahorka M, Jerliu N, Ramadani Q, Fota N, Merten S. Perceived barriers to physical activity behaviour among patients with diabetes and hypertension in Kosovo: a qualitative study. BMC Prim Care. 2022 Sep 30;23(1):257. doi: 10.1186/s12875-022-01866-w. PMID 36180857
- [Background] British Heart Foundation (2015). Cardiovascular Disease Statistics 2015: British Heart Foundation Centre on Population Approaches. Available from: https://www.bhf.org.uk/informationsupport/publications/statistics/cvd-stats-2015.
- See also: National Institute for Health and Care Excellence [NICE] (2019). Hypertension in adults: diagnosis and management — https://www.nice.org.uk/guidance/ng136/chapter/Recommendations#treating-and-monitoring-hypertension
- See also: Institute for Health Metrics and Evaluation (IHME). Global Burden of Disease 2021: Findings from the GBD 2021 Study — https://www.healthdata.org/sites/default/files/2024-05/GBD_2021_Booklet_FINAL_2024.05.16.pdf
- See also: Public Health England (2018). Tackling high blood pressure: an update — https://assets.publishing.service.gov.uk/media/5a81d95940f0b62305b91227/Tackling_high_blood_pressure_an_update.pdf